CLINICAL TRIAL: NCT01457872
Title: Malmö Treatment Referral and Intervention Study
Acronym: MATRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MATRIS
Record Dates: First submitted 2011-10-18; First posted 2011-10-24 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Heroin Addiction; Substance Use Disorders
Keywords: Heroin addiction; Substance use disorders; Substitution treatment; Syringe exchange
MeSH Terms: conditions — Heroin Dependence; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength-based case management (Experimental): Case management plus referral (vs referral-only)
  Interventions: Behavioral: Strength-based case management
- Referral only (Active Comparator): Referral only (no case management intervention)
  Interventions: Behavioral: Control condition - referral only

INTERVENTIONS:
Behavioral: Strength-based case management — Strength-based case management
  Arms: Strength-based case management
Behavioral: Control condition - referral only — Referral only
  Arms: Referral only

SUMMARY:
This study aims to study and implement active referral of heroin users from a syringe exchange programme to evidence-based treatment for heroin addiction. Patients are randomized to either a strength-based case management intervention or a control group, while both groups receive referral to medical investigation for inclusion in substitution treatment for heroin addiction. The hypothesis is that syringe exchange can be used for referral to effective treatment, and that a strength-based intervention can increase the number of patients who are successfully referred and enter treatment.

DETAILED DESCRIPTION:
Patients attending the syringe exchange programme of Malmö, Sweden, and who are using heroin as their primary drug of abuse and who live in the catchment area of Malmö Addiction Centre, will be addressed, and patients willing to participate will undergo a baseline interview and will be referred to medical examination for decision to start substitution treatment to treat heroin dependence. Half of patients will be randomized to a strength-based case management intervention, hypothesized to facilitate treatment entry, and half of patients will be randomized to a control condition involving only referral.

The study will measure the number of patients who successfully accept referral and initiate substitution treatment for heroin dependence, comparing patients in intervention arm to patients in the control condition (RCT design). Also, as a secondary outcome measure, retention and treatment outcome (substance use and clinical characteristics) will be compared between the two groups. In addition, this study will enable a number of sub-analyses aiming to increase knowledge about heroin addicts' detailed substance use pattern and clinical characteristics. Patients will be followed with respect to retention, substance use and clinical picture for three years.

ELIGIBILITY:
Inclusion Criteria:

* Registered at syringe exchange programme of Malmö
* Primary drug heroin
* Heroin dependence
* Living in catchment area for substitution treatment of Addiction Centre Malmö

Exclusion Criteria:

* Inability to understand consent and information
* Unstable psychiatric condition making treatment regulations impossible
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Treatment entry in substitution treatment at two time points - directly after referral and after up to 3 months | At medical examination after 10 days, and subsequently for up to 3 months
  Percentage of patients successfully referred for examination and start of substitution treatment. This is measured at two time points, at 10 days post-referral when the medical examination is carried out (the percentage of patients who successfully show up) and subsequently the patients will be followed up to three months post-referral with respect to actual initiation of medication.

SECONDARY OUTCOMES:
Retention and treatment outcome in substitution treatment | 3, 6, 12, 24, 26 months
  Percentage of patients remaining in treatment. Treatment outcome including decrease in substance use and improvement in clinical picture.

CONTACTS AND LOCATIONS:
Locations (1):
- Malmö Addiction Centre, Malmö University Hospital entrance 90, Malmo, Sweden